CLINICAL TRIAL: NCT04207931
Title: Treatment Results for Patients With Central Centrifugal Cicatricial Alopecia (CCCA): a Multicenter Prospective Study
Acronym: CCCA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: The Skin of Color Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00043796
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Central Centrifugal Cicatricial Alopecia (CCCA)
Keywords: alopecia; Hair loss; Female hair loss; Minoxidil; Topical Steroid
MeSH Terms: conditions — Alopecia | interventions — Clobetasol; betamethasone-17,21-dipropionate; Fluocinonide; Triamcinolone Acetonide; Doxycycline; Minoxidil

STUDY DESIGN:
Intervention Model Description: Treatment groups that patients will be randomized to include 1) topical steroid plus oral antibiotic group, and topical minoxidil after 8 months 2) topical steroid plus intralesional steroid group and topical minoxidil after 8 months.
Who Masked: Outcomes Assessor
Masking Description: To help ensure subject privacy and confidentiality, only a unique study identifier will appear on the data collection form. The data collected will be stored on the Research Electronic Database CaptureTM with access limited to designated study personnel.
  Blinded investigators from Wake Forest Baptist Department of Dermatology will later review photographs of each subject taken at baseline and at month 18 and will assign severity scores to the photographs based on the Central Scalp Alopecia Scale. These investigators will not know when each photograph was taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Topical steroid plus oral antibiotic group (Active Comparator): Participants in this group receive topical steroid (class I-II applied once daily) plus oral antibiotic group (doxycyline 100 mg twice daily for 6 months), and then topical minoxidil (5% solution or foam) after 8 months of treatment.
  Interventions: Drug: Topical steroid class I-II; Drug: Doxycyline; Drug: Minoxidil
- Topical steroid plus intralesional steroid injection group (Active Comparator): Participants in this group receive topical steroid (class I-II applied once daily) plus intralesional steroid group (7.5mg/cc of kenaolog, max dose of 3 cc), and then topical minoxidil (5% solution or foam) after 8 months of treatment
  Interventions: Drug: Topical steroid class I-II; Drug: Triamcinolone Acetonide; Drug: Minoxidil

INTERVENTIONS:
Drug: Topical steroid class I-II — applied once daily - 18 month duration of the study
  Other Names: Clobetasol, Betamethasone Dipropionate, or Fluocinonide
Drug: Triamcinolone Acetonide — Intralesional Steroid Injection, 7.5mg/cc. max dose of 3 cc. Scalp injections will be administered every 6-8 weeks, for a total of 8 injections.
  Other Names: Kenaolog
  Arms: Topical steroid plus intralesional steroid injection group
Drug: Doxycyline — oral antibiotic twice daily for 6 months
  Other Names: Doxy-100; Targadox; Oracea
  Arms: Topical steroid plus oral antibiotic group
Drug: Minoxidil — 5% solution or foam started after month 8
  Other Names: Rogaine

SUMMARY:
The objective of this study is to examine photos of CCCA patients taken before and after treatment to compare treatment outcomes between different treatment groups

DETAILED DESCRIPTION:
Treatment groups that patients will be randomized to include 1) topical steroid plus oral antibiotic group, and topical minoxidil after 8 months 2) topical steroid plus intralesional steroid group and topical minoxidil after 8 months. Both these regimens are used as the first-line treatments by clinicians. The objective of this study is to examine photos of CCCA patients taken before and after treatment to compare treatment outcomes between different treatment groups.

In this study, the investigators are looking to determine how standard treatment affects the outcome of central centrifugal cicatricial alopecia; to determine if topical steroid with With Doxycycline has better outcome than topical steroids with intralesional steroids in central centrifugal cicatricial alopecia, and to determine how the addition of topical minoxidil as a treatment changes the outcome of central centrifugal cicatricial alopecia.

ELIGIBILITY:
Inclusion Criteria:

* African-American women, ages 18-60 years old
* with a clinical diagnosis and biopsy-proven CCCA, with Central Scalp Alopecia Scale severity 1 through 4 will be included in this study
* These subjects will be seen and treated in Wake Forest Baptist Health Dermatology Outpatient Clinic

Exclusion Criteria:

* Patients with other forms of hair loss in addition to CCCA will be excluded
* Other patients to be excluded are those with other forms of inflammatory scalp disease (with the exception of mild seborrheic dermatitis)
* patients who have had topical treatment for CCCA within the past 4 months (including topical steroids, topical minoxidil, or any other topical hair regrowth medication)
* patients who have been on a long-term oral antibiotics for hair loss within the past year
* patients who have undergone more than two rounds of intralesional steroid injections to the scalp in the past one year.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — African-American women
Enrollment: 250 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Central Scalp Alopecia Photographic Scale in African American Women | baseline
  Photographs of the subject's scalp will be taken at baseline. This instrument is a 6-point scale that includes gradations in hair loss from normal (0) to bald scalp (5). Higher numbers denote greater hair loss.
Central Scalp Alopecia Photographic Scale in African American Women | Visit 4, Month 6
  This instrument is a 6-point scale that includes gradations in hair loss from normal (0) to bald scalp (5). Higher numbers denote greater hair loss.

SECONDARY OUTCOMES:
Hair Loss Questionnaire | Baseline, Visit 4, Month 6; Visit 7, Month 12; and Visit 9, Month 18-20
  Questionnaire gathers the epidemiologic data about the patient's hair loss, family history of hair loss, what treatments have been tried in the past, and hair care practices.
  There is no range and/or direction as this questionnaire is used to gather descriptive data.
Dermatology Life Quality Index (DLQI) | Visit 4, Month 6; Visit 7, Month 12; and Visit 9, Month 18-20
  Questionnaire measures how CCCA and the symptoms associated have affected daily activities over the past week. A 5-point scale is used. It ranges from 'Very Much' to 'Not Relevant' with 'Very Much' meaning that it negatively affects their daily living and quality of life and 'Not Relevant' meaning that it has no effect on their daily living and quality of life.
Last Year Dermatology Life Quality Index (LYDLQI) | Baseline
  Questionnaire measures how CCCA and the symptoms associated have affected daily activities over the past year. A 5-point scale is used. It ranges from 'Very Much' to 'Not Relevant' with 'Very Much' meaning that it negatively affects their daily living and quality of life and 'Not Relevant' meaning that it has no effect on their daily living and quality of life.
Central Scalp Alopecia Photographic Scale in African American Women | Visit 7, Month 12; Visit 9, Month 18-20
  This instrument is a 6-point scale that includes gradations in hair loss from normal (0) to bald scalp (5). Higher numbers denote greater hair loss.

CONTACTS AND LOCATIONS:
Overall Officials: Amy J McMichael, MD, Principal Investigator — Wake Forest Baptist Health Department of Dermatology
Locations (1):
- Wake Forest Baptist Health Department of Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sperling LC, Sau P. The follicular degeneration syndrome in black patients. 'Hot comb alopecia' revisited and revised. Arch Dermatol. 1992 Jan;128(1):68-74. PMID 1739290
- [Background] Bin Saif GA, Ericson ME, Yosipovitch G. The itchy scalp--scratching for an explanation. Exp Dermatol. 2011 Dec;20(12):959-68. doi: 10.1111/j.1600-0625.2011.01389.x. PMID 22092575